CLINICAL TRIAL: NCT05980221
Title: The Development of a Metabolomic Test to Diagnose and Quantify Pancreatic Exocrine Insufficiency (The DETECTION Study)
Acronym: DETECTION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Collaborators: Pancreatic Cancer UK (Other)
Responsible Party: Principal Investigator, Keith John Roberts, Consultant HPB and transplant surgeon, University Hospital Birmingham NHS Foundation Trust
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: RRK6813
Record Dates: First submitted 2023-05-31; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Pancreatic Exocrine Insufficiency
Keywords: exocrine insufficiency; pancreatic cancer; metabolomics; metabolites; chronic pancreatitis; cystic fibrosis
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Pancreatic Neoplasms; Pancreatitis, Chronic; Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Investigating the metabolome of patients with PEI in the fasted and fed state. Prospective, single centre, observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pancreatic cancer (main cohort) (Other): investigation of PEI and the metabolome of patients with pancreatic cancer in the fed and fasted state
  Interventions: Diagnostic Test: Metabolomics; Diagnostic Test: 13C MTGT
- Sub-study cohorts: Chronic pancreatitis, cystic fibrosis, NET patients on SSAs (Other): investigation of PEI and the metabolome of patients with other causes of PEI in the fed and fasted state
  Interventions: Diagnostic Test: Metabolomics; Diagnostic Test: 13C MTGT
- Dosing arm (Other): Investigation metabolome of patients pre and post initiation of PERT as part of their PEI care
  Interventions: Diagnostic Test: Metabolomics; Diagnostic Test: 13C MTGT

INTERVENTIONS:
Diagnostic Test: Metabolomics — Plasma samples taken for the investigation of the metabolome
Diagnostic Test: 13C MTGT — sequential breath samples taken for investigation of PEI (reference test)
  Other Names: 13C MTG breath test

SUMMARY:
DETECTION. The development of a metabolomic test to diagnose and quantify pancreatic exocrine insufficiency.

DETAILED DESCRIPTION:
Pancreatic exocrine insufficiency (PEI) is prevalent and progressive among patients with pancreatic cancer, treatment with pancreatic enzyme replacement therapy (PERT) has been proven to reduce gastrointestinal symptoms, improve quality of life and survival and is therefore recommended in NICE guidelines. Despite this, most patients with PEI do not receive PERT.

One cause for under treatment is lack of a well-tolerated and accurate diagnostic test that can provide quick results. The current, most widely used test, the faecal elastase stool test, has low accuracy, particularly after surgery, and results take several days. Furthermore, the test cannot help with dosing of PERT.

Metabolomics can be used to quantify metabolites in blood. These metabolites are directly influenced by normal digestion and absorption of food, for example blood lipid levels are very different in the fed and fasted states. This program of work will give a standard meal to healthy controls and patients with PEI and screen their blood before and after a test meal. Differences in the metabolic profile will be used to develop a 'fingerprint' of PEI based upon one metabolite or a combination of metabolites.

The ultimate goal is to develop a simple blood test that can be used outside of specialist centres that is acceptable to patients, can accurately diagnose PEI and can guide treatment with PERT.

This body of work aims to investigate the metabolome of patients with PEI (of different causes), PEI will be defined in the different cohorts by a multimodel approach with the 13C MTGT as primary reference test and FE-1 and PEI-Q used as supporting tests.

A test meal will be given to fasted participants alongside baseline blood samples and breath samples. Patients will then have blood and breath taken hourly for 6 hours. Blood samples will be spun and frozen for batch metabolomic analysis.

ELIGIBILITY:
Inclusion Criteria: (for main pancreatic cancer cohort)

* PDAC
* PEI (as defined by breath test)
* Tolerating oral diet Inclusion Criteria: (for CF cohort)
* CF
* PEI (as defined by breath test)
* Tolerating oral diet Inclusion Criteria: (for CP cohort)
* CP
* PEI (as defined by breath test)
* Tolerating oral diet

Exclusion Criteria (all arms):

* No other GI conditions
* For each arm no evidence of the other arm conditions
* For health controls, no history of CP, CF or pancreatic cancer
* No GI surgery (except pancreatic resection in the pancreatic cancer cohort)
* Unable to consent
* Unable to travel to UHB for testing
* Prognosis < 2months
* Performance status 2+

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Metabolome | 1 year after study completion
  metabolomic fingerprint of patient with PEI in the fed and fasted state Bloods are taken in the fed and fasted state, after centrifugation, the plasma is then frozen at -80. Samples will then be analysed using untargeted liquid chromatography mass spectrometry, after which the raw data will be processed using the open-source software XCMS. The resultant metabolite features in the samples will be compared between healthy and diseased (PEI) cohorts to identify features specific to exocrine insufficiency.

SECONDARY OUTCOMES:
PEI status using 13CMTGT in comparison to the metabolome | 1 year after study completion
  breath test (13CMTGT). 13C labelled fatty test meal ingested, exhaled breath samples eveyr hour up to 6 hours, the cumulative percent dose of 13C recovered will then be used as a marker for PEI, diagnostic under 29%
PEI status using FE-1 in comparison to the metabolome | 1 year after study completion
  FE-1. Faecal elastase, diagnostic <200
PEI status using PEIQ in comparison to the metabolome | 1 year after study completion
  PEI-Q: Pancreatic exocrine insufficiency questionnaire (symptomatic assessment of PEI). >1.8 severe PEI, 1.4-1.8 moderate PEI, 0.6-1.4 mild PEI
Response of the fed and fasted metabolome to PERT | 1 year after study completion
  Investigation of the metabolome in response to PERT low dose and high dose. The metabolomic profile indicative of PEI will then be assessed in a repeat cohort of patients that reattend twice on low dose and then high dose PERT. Bloods will be taken as for the main trial, in the fed and fasted state and the metabolomic profile (determined by the main cohort) will assessed using targeted liquid chromatography mass spectrometry to investigate whether it is altered by PERT (pancreatic exocrine replacement therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Roberts, PhD, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, United Kingdom